CLINICAL TRIAL: NCT01583907
Title: Nutrition in Children With Food Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: RBC-100789; 100789 (Other: DEPARTMENT OF PEDIATRICS UNIVERSITY OF NAPLES FEDERICO II)
Record Dates: First submitted 2012-04-05; First posted 2012-04-24 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Food Allergy
Keywords: cow's milk allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sampling to measure laboratory parameters useful to asses nutritional status
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- different dietotherapy strategies

SUMMARY:
The investigators aim to asses the effect of dieto-therapy and of nutritional counseling on the nutritional status, body growth and tolerance acquisition in children with cow's milk allergy.

DETAILED DESCRIPTION:
Prospective controlled study including patients with cow's milk allergy(6-36 months of age.During the first examination, the diagnosis will be assessed by pediatricians with great experience in food allergy, checking that the patient had undergone a standardized procedure. All cases with an unclear diagnosis of FA (i.e., lack of careful medical history, laboratory studies, and oral food challenge) or on incorrect exclusion diet (i.e., assumption of at least traces of the food allergen) will be excluded. Children with a positive history for prematurity, systemic diseases, renal failure, neurological impairment, active tuberculosis, autoimmune diseases, immunodeficiency, chronic inflammatory bowel diseases, celiac disease, cystic fibrosis, metabolic or endocrine diseases, malignancy and malformation of the gastrointestinal or the urinary tract will be also excluded. The history of each patient will be evaluated and the results of FA screening tests (i.e., skin prick tests and atopy patch tests) and of oral food challenge, together with all demographic and clinical information will be registered into a specific clinical chart. At enrolment (T0), after 2 (T1),4 (T2), 6(T3)and 12 months (T4) weight, length or height and head circumference were measured by experienced nurse unaware of the study aims using standardized procedures. The anthropometric indices (z-score for weight, z-score for length/height, z-score for head circumference) will be also evaluated for all study subjects. Anthropometric measurements will be compared with the Euro-Growth References Charts. At the end of the first visit the parents of all children taking part in the study will be asked to fill a 3-day diet record report in a form of a printed chart. Written informed consent will be obtained from parents of each child enrolled in the study.

Nutritional counseling Enrolled subjects will be evaluated by registered dieticians with a wide experience in pediatric FA, blinded to the study aims, assessing the results of the 3-day diary dietary intake at enrollment (T0), at 6 months (T3) and 12 months (T4). All diaries will be collected and analyzed using a specific software based on the Italian food composition tables. The dieticians will evaluate the results of the 3-day diary and will give information to the parents about issues potentially arising during dietary elimination and on how to replace the allergen in the diet with alternative food items equivalent on the nutritional standpoint according to specific dietary recommended intake (DRI) for Italian children for age and sex .The nutritional counseling will be also focused on feeding behaviors, selection pleasant food and children preferences. No nutritional support products will be prescribed. This is the standard procedure in the management of FA in the centers involved in the study.

Laboratory measurements At the enrollment and after 6 months (T3) after nutritional intervention a venous blood sample will be collected from children with FA on elimination diet. The following laboratory measurements will be analyzed through standardized procedures: hemoglobin, albumin, total cholesterol, triglycerides, calcium, phosphorus, and zinc.

To investigate the patients rate of tolerance acquisition after 12 months of exclusion diet an oral food challenge (OFC) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients 6-36 months of age with a suspected FA

Exclusion Criteria:

* Unconfirmed diagnosis of FA
* Prematurity
* Systemic disease
* Renal failure
* Neurological impairment
* Active tuberculosis
* Autoimmune diseases
* Immunodeficiency
* Chronic inflammatory bowel diseases
* Celiac disease
* Cystic fibrosis
* Metabolic or endocrine diseases
* Malignancy
* Malformation of the gastrointestinal or the urinary tract

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with a sure diagnosis of food allergy
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in anthropometric indices after dieto-therapy intervention and nutritional counseling in children with cow's milk allergy | 1 year
  Anthropometric indices (z-score for weight, length and head circumference) will be collected at the enrolment (T0) and after 2 (T1), 4 (T2) and 6 months (T3) by experienced nurse unaware to of the study aims. Dietary intake will be assessed by a 3-day diary at T0 and at T3. The nutrient intake will be analyzed using a specific software. The following laboratory measurements will be also analyzed at T0 and at T3: haemoglobin, albumin, total cholesterol, triglycerides, calcium, phosphorus, zinc, fatty acids.

SECONDARY OUTCOMES:
Change in nutritional status after dieto-therapy intervention and nutritional counseling in children with cow's milk allergy | 1 year
  Dietary intake will be assessed by a 3-day diary at T0 and at T3. The nutrient intake will be analyzed using a specific software. The following laboratory measurements will be also analyzed at T0 and at T3: haemoglobin, albumin, total cholesterol, triglycerides, calcium, phosphorus, zinc, fatty acids.
Change in time of tolerance acquisition after dieto-therapy intervention in children with cow's milk allergy. | 1 year
  After 12 months of dietotherapy with different formulas tolerance acquisition will be investigated performing a double blind placebo controlled oral food challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- university of naples federico II, Naples, Naples, Italy